CLINICAL TRIAL: NCT06352983
Title: Monolithic- and Partially Veneered High-translucent Zirconium Dioxide (YSZ), a 4-year Follow-up of a Multicenter Prospective, Randomized Controlled Trial on Posterior FDPs.
Brief Title: Zirconium Dioxide Fixed Dental Prosthesis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014/11
Record Dates: First submitted 2024-03-20; First posted 2024-04-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Missing Teeth
Keywords: dental ceramics; zirconium dioxide; randomized controlled trial; monolithic; FDP
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both participant, care providers, dental technicians and the investigator are blinded in the process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Veneered high-translucent zirconium dioxide fixed dental prosthesis (Experimental): Core material: high translucent zirconium dioxide (BruxZir, Glidewell, Newport Beach, Canada) Buccal veneer: porcelain (GC initial Zr, GC Corporation, Tokyo, Japan).
  Interventions: Procedure: Fixed dental prosthesis
- Monolithic high-translucent zirconium dioxide fixed dental prosthesis (Active Comparator): High translucent zirconium dioxide (BruxZir, Glidewell, Newport Beach, Canada)
  Interventions: Procedure: Fixed dental prosthesis

INTERVENTIONS:
Procedure: Fixed dental prosthesis — Fixed dentals prosthesis made out of high translucent zirconium dioxide with or without a porcelain veneer.

SUMMARY:
The purpose of this clinical trial is to evaluate and compare bridges to replace one or two missing teeth in the mouth. The bridges will be made of two variants of ceramic material. We will evaluate the bridges for up to five years regarding technical and biological complications.

DETAILED DESCRIPTION:
Purpose:

The purpose of this prospective randomized double blinded clinical trial is to systematically evaluate and compare the long-term durability of monolithic zirconium dioxide and veneered zirconium dioxide based 3-, 4- or 5-unit bridges in the posterior dentition over time. The durability will be evaluated by recording technical and biological complications.

Background:

Fixed dental prosthesis (FDP) therapy is a common therapy. Usually the FDPs are made by combining a metal frame with a veneer to give the body a more tooth-like appearance, known as porcelain-fused-to-metal.

For 20 years we have used ceramic frames as an alternative to metal, since it has better biological and aesthetic properties. A common complication with these newer materials, however, is that the porcelain veneer debonds from the substructure, which sometimes leads to a need for remaking the FDP.

Zirconium dioxide or yttria stabilized tetragonal polycrystalline zirconium dioxide (Y-TZP), is an oxide ceramic with excellent characteristics such as high strength and biocompatibility. We currently use this ceramic routinely in dentistry for the production of both crowns and FDPs. It is now a well-documented and reliable material.

The monolithic restorations, that is Y-TZP without veneer, have been developed over the past few years. The former core materials in Y-TZP were opaque white-colored but have recently undergone development to become much more esthetic by increased translucency and improving staining techniques, without losing strength. By using only the strong oxide ceramic throughout we can obtain strong materials that have good biological properties, but without the risk of porcelain veneering fractures.

Laboratory studies evaluating crown therapy have shown very good results regarding these monolithic materials, but clinical trials on FDPs are missing. The long-term clinical studies on FDPs available concern veneered Y-TZP which have achieved acceptable results with good survival rate but with some complications in the form of veneer fractures. The veneering technique and materials for Y-TZP FDPs have since been developed to decrease the risk of chip-off fractures and recent publications show promising results. The aim of this study is therefore to compare survival and complications rates of Y-TZP FDPs with veneer and without veneer, monolithic, respectively.

Question:

The null hypothesis for this study is that monolithic Y-TZP based FDPs will perform equivalent to the veneered Y-TZP based FDPs when used for constructions in the posterior dentition.

Study population:

Patients for the study will be recruited within the daily dental care operations at clinics in Public and Private Dental Services.

Study method and randomization:

Included patients will undergo treatment in the form of preparation of the teeth and an impression taken for FDP therapy. The dentist does not know which of the two different FDP materials his patient will receive. The dental laboratory will receive a requisition from the dentist with a code number. This code number is randomized to one of the two materials to be investigated. Half of the patients will get a veneered zirconia based FDP while the other half receives a monolithic zirconia based. The finished FDP will then be cemented in the same way regardless of material. Method of treatment, FDP materials and cementation is performed according to a standardized protocol used routinely in dentistry.

Evaluation methods:

The evaluation is done by recording technical and biological complications. The examination is conducted by intraoral inspection and photo documentation and is performed by dentists not involved in the performed treatments.

Quality control and reporting:

Will be published in a scientific journal.

ELIGIBILITY:
Inclusion Criteria:

Patients who needed an FDP replacing one or two missing teeth in the posterior dentition (premolars and/or molars).

Exclusion Criteria:

High caries activity Active periodontal disease Previously known history of repeated fractures of filings and/or reconstructions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Fractures | 4 years; From cementation of the fixed dental prosthesis up to the final evaluation.
  Minor or major fractures of the fixed dental prosthesis material
De-bonding | 4 years; From cementation of the fixed dental prosthesis up to the final evaluation.
  Loss of retention of the fixed dental prosthesis.

SECONDARY OUTCOMES:
Caries | 4 years; From cementation of the fixed dental prosthesis to the final evaluation.
  Biological complication, presence of caries around the fixed dental prosthesis.
Endodontic | 4 years; From cementation of the fixed dental prosthesis to the final evaluation.
  Biological complication, if there had been a need of endodontic treatment during the evaluation period.
Function | 4 years; From cementation of the fixed dental prosthesis to the final evaluation.
  Patient-reported outcome, how the patient evaluate the function of the restoration. Modified interval scale.
Esthetics | 4 years. From cementation of the fixed dental prosthesis to the final evaluation.
  Patient-reported outcome, how the patient evaluate the esthetics of the restoration.Modified interval scale.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Gardell, Principal Investigator — Malmo university
Locations (1):
- Malmo university, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
The study began enrolling patients before January 1 2019.